CLINICAL TRIAL: NCT04320147
Title: MR-target Biopsy vs. TRUS-biopsy in Men With Suspicious Prostate Cancer: A Paired Cohort Study
Brief Title: MR-target Biopsy vs. TRUS-biopsy in Men With Suspicious Prostate Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Asan Medical Center (Other)
Collaborators: Bumjin Lim (Unknown); Dalsan Yoo (Unknown); Hyung Keun Park (Unknown); Jun Hyuk Hong (Unknown); Hanjong Ahn (Unknown); Choung-Soo Kim (Unknown); Kye Jin Park (Unknown); Mi-Hyun Kim (Unknown); Jeong Kon Kim (Unknown)
Responsible Party: Principal Investigator, In Gab Jeong, Professor, Department of Urology, Asan Medical Center, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MRphI_AMC01
Record Dates: First submitted 2020-03-19; First posted 2020-03-24 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; MR-target Biopsy; Artemis
MeSH Terms: conditions — Prostatic Neoplasms; Severe combined immunodeficiency with sensitivity to ionizing radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- MRI tartget biopsy (Experimental): 1. MR-targeted biopsy using Artemis device fusion of MRI and ultrasound images would be performed. MR targeted biopsy would be performed by radiologist.
  2. Next conventional ultrasound-guided 12-core systematic biopsy would be performed by urologist. This portion will be performed without information of the MRI report.
  Interventions: Device: Artemia

INTERVENTIONS:
Device: Artemia — Before prostate biopsy, all patients be preceded by mpMRI.MR-targeted biopsy using Artemis device fusion of MRI and ultrasound images would be performed. MR targeted biopsy would be performed by radiologist.

SUMMARY:
This paired cohort blinded trial aims to assess the detection rate of clinically significant cancer of MRI-targeted biopsy compared to standard 12-core TRUS biopsy in men referred with clinical suspicion of prostate cancer who have had no prior prostate biopsy. The investigators hypothesize that additional MRI-targeted biopsy will detect more clinically significant cancers than standard TRUS biopsy.

Main objective: To compare MR-target vs. standard 12-cores TRUS-biopsy for the diagnosis of clinically significant prostate cancer.

DETAILED DESCRIPTION:
Before prostate biopsy, all patients be preceded by mpMRI. The mpMRI is read by an experienced radiologist according to the PI-RADS version 2 scoring system. PI-RADS scoring system is used to assign a degree of doubt prostate cancer. Depending on the PI-RADS score, MR targeted biopsy is determined.

1. MR-targeted biopsy using Artemis device fusion of MRI and ultrasound images would be performed. MR targeted biopsy would be performed by radiologist.
2. Next conventional ultrasound-guided 12-core systematic biopsy would be performed by urologist. This portion will be performed without information of the MRI report.

ELIGIBILITY:
Inclusion Criteria:

* 1. Men undergoing a first-time prostate biopsy to rule out cancer
* 2. Serum PSA ≥3ng/mL, ≤20ng/mL
* 3. Age≥50 years, ≤80 years
* 4. Clinical stage ≤T2c
* 5. Patients must be able to provide written informed consent.

Exclusion Criteria:

* 1. Patients has any prior needle biopsy of the prostate
* 2. Patients has a prior history of prostate cancer
* 3. Patients has a prior history of pelvic radiation therapy or androgen deprivation therapy
* 4. Patients has a prior history of BPH operation
* 5. Patient with uncorrectable coagulopathies
* 6. Unable to tolerate a TRUS guided biopsy.
* 7. Patients had 5-alpha reductase inhibitor in the past six months.
* 8. The patient has had a urinary tract infection or acute prostatitis in the last three months.
* 9. Any contraindication to MRI (severe claustrophobia, pacemaker, MRI-incompatible prosthesis, eGFR ≤50mls/min)

Ages: 50 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2020-03-23 (Estimated); Primary Completion 2021-04-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of clinically significant prostate cancer (≥Gleason score 3+4) | 2 week after the procedure

SECONDARY OUTCOMES:
Proportion of clinically insignificant prostate cancer (Gleason score 6) | 2 week after the procedure
Proportion of men in whom mpMRI score (PI-RADS) for suspicion of clinically significant cancer was 3, 4 or 5 | 2 week after the procedure
Correlation of prostate health index (Phi), phi density and MRI fusion Bx in predicting clinically significant prostate cancer | 2 week after the procedure
Cancer core length of the most involved biopsy core (maximum cancer core length, mm) | 2 week after the procedure
Proportion of men who go on to definitive local treatment or systemic treatment | 2 week after the procedure
Proportion of Gleason grade upgrading in men undergoing radical prostatectomy | 2 week after the surgery
Adverse events of post-biopsy (pain, infection, bleeding etc.) | 2 week after the procedure
Inter-observer variability among radiologists | 2 week after the procedure

CONTACTS AND LOCATIONS:
Overall Officials: In Gab Jeong, MD, PhD, Study Chair — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No